CLINICAL TRIAL: NCT01169142
Title: A Pilot Study of Vitamin D Supplementation in Bronx Psychiatric Patients
Brief Title: Study of Vitamin D in the Severely Mentally Ill
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bronx Psychiatric Center (Other Government)
Responsible Party: Principal Investigator, Nigel Bark MD, Director of Scizhophrenia Research, Bronx Psychiatric Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BPCIRB0804
Record Dates: First submitted 2010-07-21; First posted 2010-07-26 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Vitamin D; Schizophrenia; Severely Mentally Ill
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate Vitamin D3 (Active Comparator): Will start Vitamin D3 immediately
  Interventions: Dietary Supplement: Vitamin D3
- Three month delay (Active Comparator): Half the subjects will be delayed three months (but evaluated) before getting Vitamin D3. (If the level is very low they will start immediately)
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — 50,000 units of Vitamin D3 weekly
  Other Names: Cholecalciferol
  Arms: Three month delay
Dietary Supplement: Vitamin D3 — Vitamin D3 50,000 units weekly
  Other Names: Cholecalciferol
  Arms: Immediate Vitamin D3

SUMMARY:
Supplementation of Vitamin D in those with low levels will increase the level and result in some improvement in health and psychopathology measures.

DETAILED DESCRIPTION:
Subjects with levels of Vitamin D between 7ng/ml and 30ng/ml will, after signing consent forms, be randomly assigned to either start immediately on Vitamin D for three months or to start after a delay of three months. Those with levels below 7gn/ml will start immediately. All will be evaluated monthly with blood tests, PANSS, movement disorder ratings and information on health and progress from the clinical chart.

ELIGIBILITY:
Inclusion Criteria:

* Age 19-70,
* Schizophrenia or Schizoaffective disorder
* stabilized but not expecting to be discharged soon
* capacity to give informed consent

Exclusion Criteria:

* acutely psychotic
* acutely medically ill
* renal insufficiency
* hypercalcemia
* hyperparathyroidism

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-01; Primary Completion 2014-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Psychopathology as measured by the PANSS | 3 months
  PANSS is being done every month

SECONDARY OUTCOMES:
movement disorder | three months
  AIMS (for tardive dyskinesia), Simpson-Angus (for Parkinsonism) and Barnes (for Akathisia) movement disorder rating scales will be completed monthly.
General Health | three months
  Measured by staff observation and reports, Labs for example glucose mg/dL, HgbA1c %A1c, Vitamin D ng/ml, calcium mg/dL, assessed monthly

CONTACTS AND LOCATIONS:
Overall Officials: NIgel Bark, MD, Principal Investigator — Bronx Psychiatric Center
Locations (1):
- Bronx Psychiatric Center, The Bronx, New York, United States